CLINICAL TRIAL: NCT02205866
Title: Incidence of Not Receptive Endometrium During the Window of Implantation as Body Mass Index by Testing ERA.
Brief Title: Incidence of Non Receptive Endometrium in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Jose Bellver, Dr. Jose Bellver, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1403-VLC-012-JB
Record Dates: First submitted 2014-07-25; First posted 2014-07-31 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Non Obese patients
  Interventions: Other: Endometrial Receptivity Array analysis of endometrial biopsy
- Group B (Experimental): Obese patients
  Interventions: Other: Endometrial Receptivity Array analysis of endometrial biopsy

INTERVENTIONS:
Other: Endometrial Receptivity Array analysis of endometrial biopsy — A biopsy of endometrium is peformed and Endometrial Receptivity Array analysis is carried out, as well as analysis of fat distribution and risk factors of Metabolic Syndrome.

SUMMARY:
This study evaluates the incidence of Non Receptive endometrium in obese infertile women compared to infertile normal weight women using Endometrial Receptivity Array (ERA) test, containing 238 genes, identifying the receptivity status of an endometrial sample and diagnosing the patient's Window of Implantation, regardless of the histological appearance of the sample. An endometrial biopsy is collected from the uterine fundus, either in a natural cycle or in a hormonal replacement therapy (HRT) cycle and the test is performed.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women: > 1 year of regular unprotected intercourse without evidence of pregnancy.
* Normal uterus by 2D/3D ultrasound scan and/or hysteroscopy
* No endometriosis
* Presence of both ovaries
* < 45 years old (in ovum donation, outcome parameters are not affected until this age in all the current published studies).

Exclusion Criteria:

* Hydrosalpinx
* Stage 3-4 endometriosis diagnosed with ultrasound, laparoscopy/ laparotomy.
* Implantation failure (≥ 4 pre-embryos of good quality transferred without pregnancy)
* Recurrent pregnancy loss (≥ 2 pregnancies biochemical / clinical)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Non Receptive Endometrium | 25 days
  To evaluate the incidence of Not Receptive endometrium in obese infertile women compared to infertile normal weight women using an adequate sample size.

SECONDARY OUTCOMES:
Distribution of fat and risk factors | 4 months
  Carry out a subanalysis concerning the distribution of central and peripheric fat and risk factors of metabolic syndrome including: Age (years); Height (m); Weight (kg) ; BMI (kg/m2); Waist (cm) ; Hip (cm); Index waist-hip ratio (WHR) waist (cm) / hip (cm); Blood pressure; insulinemia Fasting blood glucose (mmol / L); PTG ( tolerance oral glucose ) (mmol / L), Total cholesterol and fractions; Triglycerides Microalbuminuria; bA1C, HC-reactive protein.
Look for specific endometrial gene patterns. | 25 days
  Find patterns of expression of specific genes in endometrial obese women: we will by analyzing the expression of 238 genes obtained after endometrial endometrial biopsy.
Evaluate the result of assisted reproduction treatment. | 12 months
  Relate if the displacement of the WOI induced by the obesity is clinically relevant after the personalized embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bellver, MD PhD, Principal Investigator — IVI Valencia
Locations (3):
- United States (2):
  - Stamford University, Palo Alto, California
  - Baylor College of Medicine, Houston, Texas
- IVI Valencia, Valencia, Spain

REFERENCES:
- [Derived] Comstock IA, Diaz-Gimeno P, Cabanillas S, Bellver J, Sebastian-Leon P, Shah M, Schutt A, Valdes CT, Ruiz-Alonso M, Valbuena D, Simon C, Lathi RB. Does an increased body mass index affect endometrial gene expression patterns in infertile patients? A functional genomics analysis. Fertil Steril. 2017 Mar;107(3):740-748.e2. doi: 10.1016/j.fertnstert.2016.11.009. Epub 2016 Dec 2. PMID 27919438